CLINICAL TRIAL: NCT04899804
Title: Investigation of the Validity and Reliability of Core Performance and Functional Capacity Tests Applied by Tele-Assessment in Healthy Individuals
Brief Title: Validity and Reliability of Tele-Assessment Based Core Performance and Functional Capacity Tests in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Feray Güngör, Physiotherapist, Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: IUC2
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: validity; reliability; telehealth; trunk endurance; functional capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validity and Reliability Group: This study will be completed in two phases. In the first phase, the participants included in the study will be evaluated first by tele-assessment. One hour later, all assessments will be repeated face-to-face procedures by the researchers; thus, the validity of the tele-assessment method will be determined. Before the tele-assessment, participants will be informed about having a chair whose floor-to-seat height is 48 cm and tape measure. In the second phase of the study, to determine the reliability of the tele-assessment method, all tests will be applied to the previously tested participant by the same researcher one week later and at the same time of the day using only the tele-assessment method.

SUMMARY:
The COVID-19 pandemic process has created the need for social isolation and quarantine, and restrictions have occurred in access to healthcare services. In this process, the trend towards alternative methods that will provide access to health services and the need for telehealth services has increased. As a result of this, when we look at the literature, evaluation methods used in the clinical environment in physiotherapy are frequently encountered in tele-evaluation. There is a need for validity and reliability studies of these evaluation methods in terms of tele-assessment. This study was designed to determine the validity and reliability of trunk endurance and functional capacity tests applied by the tele-assessment method in healthy individuals.

DETAILED DESCRIPTION:
Tele-health has become a service whose prevalence has increased in recent years with the development of technology. Tele-health facilitates the accessibility of health services for individuals in all segments of society. Telerehabilitation, a subcomponent of telehealth, provides easy access to rehabilitation services by reducing cost, time, and distance barriers in physiotherapy. It offers physiotherapists the opportunity to observe the musculoskeletal system through physical assessment, exercise program planning, distance education, and continuous feedback of individuals. In this sense, tele-assessment has an important place within the scope of health services. As a result of the restrictions that came with the COVID-19 process, it has become difficult for individuals to access health services. With the effective use of technology to eliminate this obstacle, telehealth has become an alternative method. Tests such as curl-up, push-up, plank, and lateral bridge are frequently used to evaluate trunk endurance in healthy individuals. For functional evaluation, the timed sit and test, the timed stand up and test, the functional anterior reach test and the one-foot balance test are among the most used tests in the literature. The validity and reliability of these methods used in the face-to-face evaluation should be determined for the correct and effective tele-assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Does not have any diagnosed disease
* Volunteer
* Able to use the technology required for tele-assessment

Exclusion Criteria:

* Do not have the technology required for evaluations
* Not willing to participate in the study
* Who have a balance problem

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Curl-up | Baseline
  The Curl-Up test is used to evaluate the trunk flexor muscle strength. In the test, individuals are asked to lie on their back, bring their hips and knees to a 90º flexion position, and perform trunk flexion for 30 seconds. In our study, the result of the Curl-up test will be recorded as the number of repetitions made by individuals for 30 seconds.
Modified Push-up | Baseline
  Push-up test is used to evaluate general core muscle strength. In the test, individuals are asked to lie in the prone position, bring their hands to shoulder level, their elbows in flexion and to the side of the body, while in this position, they are asked to raise the head, shoulder and trunk with the elbows fully extended for 30 seconds. In our study, the number of repetitions performed by the subjects for 30 seconds will be recorded.
Plank | Baseline
  Plank test will be applied to evaluate general core endurance. Participants will be positioned so that their forearms and toes are on the ground and they will be asked to lift their trunk by giving weight. Participants will be informed about the correct alignment of the whole body during the test. The time in which the body's position is maintained will be recorded in seconds and the test will be terminated as soon as the position is broken.
Lateral bridge | Baseline
  The lateral bridge test is used to test the endurance of the lateral trunk muscles. n the test, the person lying on his back is asked to turn sideways on one side, place his forearm on the ground at an angle of 90º with the arm, and cross his upper arm to the opposite shoulder. The subject is asked to lift his body up on his forearm and toes while in this position and to maintain this position. In our study, with the lateral bridge test, the time that the patients stand without disturbing the movement will be recorded in seconds by means of the stopwatch, the test will be repeated twice for both sides and the best result will be evaluated.
30 seconds sit to stand test (30STS) | Baseline
  30STS is used to evaluate lower extremity functionality and dynamic balance. A chair with a hard seat which a floor-to-seat height of 48 cm will be stabilized. Participants will be asked to sit with their feet flat on the ground and their upper limbs crossed to their chest. Participants will be asked to stand up and sit for 30 seconds and the number of repetitions will be recorded.
Timed up and go test (TUG) | Baseline
  TUG is used to measure basic mobility. Time is registered from when the participant arises, walks 3 m, turns around, walks back, and sits down again. A test trial will be allowed, and two attempts will be registered.
Functional reach test (FRT) | Baseline
  FRT is an outcome measure used to assess dynamic balance in a task. In standing, the distance between the length of an outstretched arm in a maximal forward reach will be measured, while maintaining a fixed base of support.

CONTACTS AND LOCATIONS:
Overall Officials: Yıldız Analay Akbaba, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Feray Güngör, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Gungor F, Ovacik U, Ertan Harputlu O, Yekdaneh AA, Kurt I, Erturk Uzunoglu G, Polat Ilguz B, Akuzum F, Akbaba YA. Tele-assessment of core performance and functional capacity: Reliability, validity, and feasibility in healthy individuals. J Telemed Telecare. 2024 Jul;30(6):1017-1025. doi: 10.1177/1357633X221117335. Epub 2022 Aug 2. PMID 35916001